CLINICAL TRIAL: NCT05331274
Title: The Effect of Structured Pain Education on Pain and Performance Parameters in Patients With Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Ayşe Yaşar, physiotherapist, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MedipolUniversity
Record Dates: First submitted 2022-03-15; First posted 2022-04-15 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise group (Experimental): Only DYMK exercise training will be applied to the exercise group.
  Interventions: Other: exercise group
- pain training group (Experimental): In the pain training group, pain training will be applied in addition to the DYMK exercise training.
  Interventions: Other: pain training group

INTERVENTIONS:
Other: exercise group — 1 stage
  * In a sitting position, pull the leg up and extend the knee forward
  * Standing, bending forward and bending the knee
  * Supine, tucked legs
  * Maintaining spinal smoothness in crawling
  * Prone heel pull to buttock
  Stage 2
  * Prone on forearms-hands
  * Extending the supine hands to the knees
  * Rounding and hollowing the waist in crawling
  * Progressive sit-stand
  * Standing up from sitting and putting on and taking off socks
  * Reaching up while standing and maintaining the straightness of the spine
  * Squatting
  * Climbing and descending stairs
  Stage 3
  * Maintaining standing, arms forward
  * Slipping hands on the bed while standing
  * Initiating the standing throw and maintaining the position until the final interval
  * Putting on and taking off socks while standing
  * Taking weight towards the ground from a certain height
  * Picking up different weights from the ground
  * Push-pull items
  * Crossing obstacles of certain height
  * Walking a certain distance
  Arms: exercise group
Other: pain training group — The training provides participants with the opportunity to explain the central sensitization mechanism and also integrates the behavioral, psychological and environmental aspects that contribute to the persistence of pain. It is intended to teach that education reduces pain and improves endogenous pain inhibition, mental health, physical function, vitality and self-rated disability in patients with chronic pain, and reduces passive coping, kinesiophobia, and catastrophizing.
  The same exercises will be applied as the exercise group.
  Arms: pain training group

SUMMARY:
The Effect of Structured Pain Education on Pain and Performance Parameters in Patients with Chronic Low Back Pain

The aim of this study is to compare the effects of only Low Load Motor Control Exercises and Pain Education in addition to these exercises on pain, performance, disability and psychological factors, and to present a generalizable pain education in patients with chronic low back pain. We think that DYMK exercises applied together with a general Pain Education given to the patients will provide more improvement on these factors.

The patients will be divided into 2 groups, as a pain training group and an exercise group, with 20 people in each group, in a randomized controlled manner. Only DYMK exercise training will be applied to the exercise group. In the pain training group, pain training will be applied in addition to the DYMK exercise training.

As an evaluation parameter to the participants; Numerical Rating Scale, Short-Form McGill Pain Questionnaire, Pain Catastrophizing Scale, Tampa Kinesiophobia Scale, Roland-Morris Disability Questionnaire, Pain Self-Efficacy Questionnaire, Passive Lumbar Extension Test, Finger-Place Test and Physical Performance Test Battery will be applied. Patients will be evaluated before the start of the study (T0) and at the end of the study (T1).

Low Load Motor Control Exercises will be applied to people in both groups for 4 weeks, 3 days a week, during 20-30 minute sessions. In addition to the DYMK exercise training, a session of 30 to 50 minutes of Pain Training in groups of 4 to 5 people will be given to the patients included in the Pain Training group at the beginning of the exercise training and the exercise training will begin.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old
* Chronic low back pain 3 days a week and ≥ 3 months
* Absence of spinal fracture or acute disc herniation
* Absence of existing psychiatric problems and mental deficiencies
* Absence of exercise contraindications [28] [29] [30]

Exclusion Criteria:

* Being diagnosed with lumbar radiculopathy
* Pain due to tumors or infections, metastases, osteoporosis, inflammatory arthritis or fractures
* Specific medical conditions (neck or back surgery in the previous 3 years, osteoporotic vertebral fractures or rheumatological diseases)
* Chronic widespread pain syndromes (fibromyalgia or chronic fatigue syndrome)
* Receiving any other treatment for chronic low back pain during the study [28] [29] [30]

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of pain intensity on the Numerical Rating Scale at 3 weeks | baseline and 3 weeks
  It is an 11-point unidimensional measure of pain intensity. It is a segmented numerical version of the Visual Analog Scale (VAS), in which participants select an integer (0-10 integer) that best reflects the intensity of their pain. 0 represents no pain and 10 represents worst pain.
Change from baseline in the multidimensional measure of pain on the Short-Form McGill Pain Questionnaire at 3 weeks | baseline and 3 weeks
  A multidimensional measure of pain. It consists of 2 subscales: 1) a sensory subscale consisting of 11 words or items, and 2) an emotional subscale consisting of 4 items rated on the intensity scale (0= none, 1= mild, 2= moderate, and 3= severe). It also includes 1 item for current pain intensity and 1 item for 10 cm Visual Analog Scale for mean pain.
Change from baseline in assessing feelings, thoughts, and emotions related to pain and disaster on the Pain Catastrophizing Scale at 3 weeks | baseline and 3 weeks
  It is used to assess the patient's feelings, thoughts, and feelings about pain and disaster. It is a self-administered questionnaire with 13 items and 3 subscales: helplessness, magnification, and rumination. A 5-point scale is used for each item, with higher values representing greater destruction. The scores of each item are added to determine the subscales and the total score is calculated with the sum of all items. Scores range from 0 to 52 points.
Change from baseline in measuring fear of movement and (re)injury on the Tampa Kinesiophobia Scale at 3 weeks | baseline and 3 weeks
  A 17-item questionnaire that measures fear of movement and (re)injury. Each question is answered on a 4-point Likert scale ranging from "strongly disagree" to "strongly agree". The total score is calculated after reversing the individual scores of items 4, 8, 12, and 16.
Change from baseline in questioning pain-related disability from low back pain on the Roland Morris Disability Questionnaire at 3 weeks | baseline and 3 weeks
  A 24-item self-reported outcome measure questioning pain-related disability from low back pain. Items are scored 0 if left blank or 1 if approved. The total score ranges from 0 to 24; higher scores represent higher pain-related disability.
Change from baseline in the patient's ability to perform a range of activities despite pain in the Pain Self-Efficacy Questionnaire at 3 weeks | baseline and 3 weeks
  A 10-item questionnaire that measures both the strength and generality of a patient's beliefs about their ability to perform a range of activities despite pain. Scores can range from 0 to 60, with higher scores indicating stronger self-efficacy beliefs.
Measuring pain intensity and disability in the Revised Graded Chronic Pain Scale at baseline | baseline
  The new scale, consisting of 6 questions, was developed as a revised version of the original scale. There is a categorical rating scheme and numerical self-assessment scores for pain intensity and disability. The first 2 questions ask the frequency of pain, how the pain affects life and work activities and evaluate the last 3 months. It is scored from 0 to 4 (0 = never to 4 = every day). Questions between 3 and 5 (PEG scale) evaluate the severity of pain in the last 7 days and are scored between 0-10 points. The third question questions the severity of the pain. Questions 4 and 5, respectively, ask how pain interferes with enjoying life and how it affects general activities. Question 6 has 2 answers (1=yes and 2=no) and asks if the person is not working or unable to work because of pain or painful condition.
Change from baseline in assessing internal factors and emotions influencing the experience of health-threatening physical injury and pain in the Pain Beliefs Questionnaire at 3 weeks | baseline and 3 weeks
  The consists of two subscales. The organic beliefs subscale (PBQ-O) questions the user about physical injury or physiological pain that threaten wellness, while the psychological pain beliefs subscale (PBQ-P) evaluates intrinsic factors and emotions affecting the pain experience that may potentially threaten wellness.
Identifying subjective neuropathic pain experience on the Pain Perception Questionnaire at baseline | baseline
  It is a symptom-based assessment tool performed by clinicians to specify the subjective neuropathic pain experience of patients.
Change from baseline in assessing overall quality of Sleep at 3 weeks | baseline and 3 weeks
  It's about the overall quality of sleep about most nights in the last 7 days. It is scored between 1 and 10. High scores represent good sleep quality.

SECONDARY OUTCOMES:
Change from baseline in detecting structural lumbar segmental instability on Passive Lumbar Extension Test at 3 weeks | baseline and 3 weeks
  It is a passive test that detects structural lumbar segmental instability. Participants are placed in a prone position and the physiotherapist then lifts both lower extremities simultaneously to a height of approximately 30 cm from the bed while keeping the knees extended and gently pulling the legs. The test is considered positive if the participant reports low back pain during testing.
Change from baseline on trunk mobility on the Finger-Place Test at 3 weeks | baseline and 3 weeks
  It is a test that provides information about trunk mobility. The participant stands upright on a 20 cm high platform, with shoes off and feet glued together. He is asked to bend forward as much as possible, fully extending his knees, arms and fingers. The vertical distance between the tip of the middle finger and the platform is measured with a flexible tape measure and expressed in centimeters. The vertical distance between the platform and the tip of the middle finger is considered positive when the participant does not reach the platform, and negative when they can go further.
Change from baseline in maintaining a neutral lumbar spine in the Physical Performance Test Battery at 3 weeks | baseline and 3 weeks
  Includes bias bridge, side bridge, Biering-Sørensen test and a motion control test battery. . All tests will be performed in standard positions. In the bias bridge, side bridge and Biering-Sørensen testing, emphasis will be placed on maintaining a neutral lumbar spine for as long as possible (seconds).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Sefakoy Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No